CLINICAL TRIAL: NCT00502489
Title: Computer Driven Management of Weaning Following Prolonged Mechanical Ventilation: a Pilot Study
Brief Title: Computer Driven Management of Weaning Following Prolonged Mechanical Ventilation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Rabin Medical Center (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 4242
Record Dates: First submitted 2007-07-15; First posted 2007-07-17 (Estimated); Last update posted 2007-07-17 (Estimated); Status verified 2007-05

CONDITIONS: Mechanical Ventilation; Weaning; Prolonged Ventilation
Keywords: prolonged mechanical ventilation; weaning;rehabilitation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: Closed-loop sytem for5 weaning from mechanical ventilation

SUMMARY:
After an episode of acute respiratory failure requiring mechanical ventilation, weaning the patient from the ventilator may be difficult. Discontinuation of ventilation is estimated to take up to 40% of the total duration of ventilatory support. Approximately two- thirds of patients can be disconnected from the ventilator after a spontaneous breathing trial. Prolongation of mechanical ventilation may increase the risk of adverse events such as infections and can increase morbidity and mortality.

Identifying weaning readiness early and reliably is therefore crucial. Weaning protocols developed to assist in identifying weaning readiness have been shown to shorten duration of mechanical ventilation, most notably the weaning period.

Closed loop knowledge-based systems serve as a continuously applied weaning process that automatically reduce ventilatory assistance according to patient ability and indicate when the patient is ready for disconnection. No data on the use of such a computer driven system (CDS) in elderly patients requiring prolonged ventilation in weaning centers (non ICU) have been reported.

The Objective of the present study is to evaluate the ability of a computer driven system to predict weaning readiness and to compare this to a physician-directed protocol. The CDS continuously adapts pressure support, gradually decreasing ventilator assistance according to patient ability, and thus indicates weaning readiness. Patients who maintain spontaneous breathing for 7 days following weaning will be considered to be successfully weaned from mechanical ventilation.

DETAILED DESCRIPTION:
Introduction.

After an episode of acute respiratory failure requiring mechanical ventilation, weaning the patient from the ventilator may be difficult. Discontinuation of ventilation is estimated to take up to 40% of the total duration of ventilatory support. Approximately two- thirds of patients can be disconnected from the ventilator after a spontaneous breathing trial. Prolongation of mechanical ventilation may increase the risk of adverse events such as infections and can increase morbidity and mortality.

Identifying weaning readiness early and reliably is therefore crucial. Weaning protocols developed to assist in identifying weaning readiness have been shown to shorten duration of mechanical ventilation, most notably the weaning period.

Closed loop knowledge-based systems serve as a continuously applied weaning process that automatically reduce ventilatory assistance according to patient ability and indicate when the patient is ready for disconnection. No data on the use of such a computer driven system (CDS) in elderly patients requiring prolonged ventilation in weaning centers (non ICU) have been reported.

Objective:

To evaluate the ability of a computer driven system to predict weaning readiness and to compare this to a physician-directed protocol. The CDS continuously adapts pressure support, gradually decreasing ventilator assistance according to patient ability, and thus indicates weaning readiness. Patients who maintain spontaneous breathing for 7 days following weaning will be considered to be successfully weaned from mechanical ventilation.

Design and setting:

A single center, randomized, controlled clinical study at the Beit Rivka regional weaning center (RWC).

Patients.

This study will be conducted at the Beit Rivka geriatric rehabilitation hospital, Petah Tikva. Written informed consent will be obtained from the patient or legal representative. The study will include 60 consecutive patients who meet all inclusion criteria after stabilization of the acute health problems that prompted admission to the referral hospital. Inclusion criteria are as follows: pressure support ventilation (PSV) for at least 48 h, plateau pressure less than 30 cmH2O, PEEP < 6 cmH2O, PaO2/FIO2 ratio > 150 or SaO2 > 94% with FIO2 < than 0.5, pCO2 <55 mm Hg for normal patients and < 65 m Hg for patients with COPD, no requirement for inotropic support, body temperature > 36.50C and < 38.50 C, stable neurological status with Glasgow Coma Score (GCS) > 6, HgB > 8 mg %, systolic blood pressure >90 mg Hg, mean arterial pressure >65 mg Hg, absence of sedative medications and availability of CDS at the time of patient admission or switching to pressure support ventilation (PSV). Patients younger than 60 or older than 85 years of age, patients on chronic ventilatory assistance at home, and patients with decision to limit life-sustaining treatments will be excluded.

Treatment group assignment will be by a sealed envelope upon admission to the hospital. Attending doctors will not be blinded as to the treatment groups.

Description of the computer driven system.

The CDS is a knowledge- based system embedded in a ventilator (EVITA XL) (15, 16, 17). It achieves three main goals. First, the CDS continuously adjusts the PSV level based on respiratory rate (RR), tidal volume (Vt) and end-tidal partial pressure of CO2 (PETCO2) acquired from the ventilator in real time and averaged over 2 min. Adjustment is such that the patient is kept within a "comfort zone" defined as a RR between 15-30 range (up to 34 within patients with neurological disorders), Vt greater than 300 ml (< 250 ml if body weight < 55 kg), and PETCO-2 less than 55 mm Hg (< 65 mmHg in patients with COPD). Second, the CDS gradually decreases ventilatory assistance by reducing PSV level after at least 30 min of stable ventilation within the comfort zone; the reduction is by 2 or 4 cm H20 depending on whether the initial level is below or above 20 cm H2O, respectively. Third, the CDS evaluates weaning readiness: when the PSV level reaches the preset minimal value (9 cm H2O in tracheotomized patients), the CDS starts an observational period, which serves as automatic spontaneous breathing trial. After uninterrupted ventilation at the minimal PSV level for 1 or 2 h (depending on whether the initial PSV level was above or below 15 cm H2O), the CDS displays a message that the patient is ready to be disconnected from the ventilator. The investigator will have perfect knowledge of the system.

Prediction of weaning. Weaning readiness as evaluated by the CDS and by the internist will be recorded daily, i.e., every morning between 10 and 11 a.m. The decision will be considered to be taken by the CDS before the physician when it was taken 1 day in advance, i.e., the preceding morning. Physicians will be aware of the PSV level delivered by the CDS and could take this level into account in their evaluation. Weaning protocols used routinely in the center recommend a daily assessment for weaning similar to that used by the CDS. Patients are declared weaned as soon as the physician or CDS predicts weaning readiness. The control group reflects the standard of care before CDS implementation. PS of 10 cm H2O or higher is set manually. After 20 min, in the absence of signs of poor tolerance, the PSV is reduced by 4 or 2 cm H20 (depending on initial PSV level > or < 20). If poor tolerance to weaning is evident, the progression of the weaning is stopped, and the patient is reassessed 20 min later for further reduction in PSV. The PSV level is decreased to 9 cm H2O. In the case of apnea, SIMV is reinstituted. If the evaluation is satisfactory, the patient is disconnected from the ventilator. The patient is closely monitored for signs of respiratory failure requiring reinstitution of mechanical ventilation, as well as for occurrence of any other complications. RWC length of stay on MV will be recorded.

Clinical characteristics including age, sex, anthropometrical data, APACHE II score, Functional Independence Measure (FIM), Mini Mental State Examination (MMSE), Geriatric Depression Scale (GDS), Mini Nutritional Assessment (MNA), temperature, ny concomitant medications, hand grip strength will be recorded.

Expired tidal volume, respiratory rate, Peak airway pressure, mean airway pressure, Compliance, Resistance, respiratory frequency to tidal volume ratio (f/Vt ), Negative Inspiratory Pressure (NIP), Maximal Inspiratory Pressure (MIP), Minute Ventilation (MV),inspiratory time will be recorded .

Other elements relevant to mechanical ventilation management include arterial blood gas estimation, the number of changes in the settings of the ventilator performed by the health care workers, the number of transitions from controlled to assisted ventilation, and the number of apnea and high pressure alarms.

The primary outcome variables will be the duration of mechanical ventilation .

Discontinuation from MV will be attempted when the primary physician judges that the patient is ready to be weaned, according to the standard criteria. Mechanical ventilation will be reinstituted in the following circumstances: respiratory rate above 35 breaths /min, P02 below 65 mm Hg with FIO2less than 0.6, ph 7.34 or less, heart rate equal to or above 1 10 beats min or Increased by 20 % or more, or if arrhythmias appear, systolic blood pressure without inotropes <90 mmHg or above 20% of usual blood pressure, uncoordinated thoraco-abdominal movements, activation of accessory muscles, agitation or depressed mental status, or excessive sweating.

A weaning trial will be considered a failure when the patient will be not tolerate the weaning trial, patients still in the use CDW at day 60 and patients requires reconnection to MV. Weaning trial will be considered successful if spontaneous breathing is sustained for more than 168 h (7 days) after disconnection from MV .

ELIGIBILITY:
Inclusion Criteria:

* Pressure support ventilation (PSV) for at least 48 h,
* Plateau pressure less than 30 cmH2O,
* PEEP < 6 cmH2O, PaO2/FIO2 ratio > 150 or SaO2 > 94% with FIO2 < than 0.5,
* pCO2 <55 mm Hg for normal patients and < 65 m Hg for patients with COPD,
* No requirement for inotropic support,
* Body temperature > 36.50C and < 38.50 C,
* Stable neurological status with Glasgow Coma Score (GCS) > 6, HgB > 8 mg %,
* Systolic blood pressure >90 mg Hg,
* Mean arterial pressure >65 mg Hg,
* Absence of sedative medications and availability of CDS at the time of patient admission or switching to pressure support ventilation (PSV).

Exclusion Criteria:

* Patients younger than 60 or older than 85 years of age,
* Patients on chronic ventilatory assistance at home; and
* Patients with decision to limit life-sustaining treatments

Ages: 60 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2007-10; Study Completion 2008-11 (Estimated)

PRIMARY OUTCOMES:
Maintenance of spontaneous breathing | 7 days

CONTACTS AND LOCATIONS:
Overall Officials: Gregory Papirov, MD, Principal Investigator — Rabin Medical Center, Beilinson Hospital, Israel